CLINICAL TRIAL: NCT07171463
Title: Evaluation of the Safety and Efficacy of Pulmonary Vein Isolation for Paroxysmal Atrial Fibrillation Using Point-by-Point Bipolar Pulsed Field Ablation Combined With Thermal Ablation of the Superior Paraseptal Parasympathetic Ganglion Region
Brief Title: Pulsed Field Ablation With Concomitant Radiofrequency Cardioneuroablation in Patients With Paroxysmal Atrial Fibrillation
Acronym: PFACNA-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Centre, Poland (Other)
Responsible Party: Principal Investigator, Łukasz Zarębski, MD, St. Joseph's Centre, Poland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12/2025/B
Record Dates: First submitted 2025-08-29; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation (Paroxysmal)
Keywords: Atrial fibrillation; Pulsed Field Ablation; Cardioneuroablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PFA with selective thermal ganglion ablation (Experimental): Participants will undergo pulmonary vein isolation using a point-by-point bipolar pulsed-field ablation. In addition, selective thermal ablation using radiofrequency energy will be performed at the anterior aspect of the right superior pulmonary vein, corresponding to the anatomical region of the superior paraseptal parasympathetic ganglion.
  Interventions: Procedure: Pulmonary Vein Isolation using Point-by-Point Bipolar Pulsed-Field Ablation; Procedure: Selective Radiofrequency Ablation of the Superior Paraseptal Parasympathetic Ganglion
- Standard PFA pulmonary vein isolation (Active Comparator): Participants will undergo pulmonary vein isolation using the same point-by-point bipolar PFA system without any additional thermal applications.
  Interventions: Procedure: Pulmonary Vein Isolation using Point-by-Point Bipolar Pulsed-Field Ablation

INTERVENTIONS:
Procedure: Pulmonary Vein Isolation using Point-by-Point Bipolar Pulsed-Field Ablation — Pulmonary vein isolation is performed via transseptal access to the left atrium using a point-by-point bipolar pulsed-field ablation catheter
Procedure: Selective Radiofrequency Ablation of the Superior Paraseptal Parasympathetic Ganglion — Targeted application of radiofrequency energy at the anterior aspect of the right superior pulmonary vein, corresponding to the anatomical location of the superior paraseptal parasympathetic ganglion.
  Arms: PFA with selective thermal ganglion ablation

SUMMARY:
Pulsed-field ablation (PFA) is a novel, non-thermal method for the treatment of atrial fibrillation (AF). It uses short, high-voltage electrical pulses to selectively ablate cardiomyocytes. PFA has demonstrated a high safety profile with reduced complication rates compared to thermal ablation.

Thermal ablation of parasympathetic ganglia during conventional pulmonary vein isolation (PVI) may improve long-term procedural outcomes by reducing AF recurrence. However, due to its non-thermal nature, PFA may not significantly affect cardiac autonomic innervation, which could be clinically relevant in vagally mediated AF or tachycardia-bradycardia syndrome.

This randomized study compares two strategies: (1) PFA-only PVI, and (2) PFA combined with selective thermal ablation (radiofrequency energy) of the superior paraseptal parasympathetic ganglion. The primary objective is to evaluate whether adjunctive thermal ablation improves clinical outcomes and reduces intraprocedural bradyarrhythmic events.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Documented paroxysmal atrial fibrillation (AF) lasting ≥30 seconds on ECG or Holter monitoring
* Willingness and ability to provide written informed consent
* Life expectancy >1 year

Exclusion Criteria:

* Persistent AF lasting >7 days or long-standing AF >1 year
* Secondary AF due to electrolyte imbalance, thyroid disease, alcohol abuse, or other non-cardiac causes
* Left atrial anteroposterior diameter ≥45 mm on transthoracic echocardiography
* Clinically significant coexisting arrhythmias other than AF
* Significant valvular heart disease or valve prosthesis
* Chronic heart failure NYHA class III/IV
* Previous AF or atrial flutter ablation
* Prior closure of atrial septal defect or left atrial appendage
* Atrial myxoma
* Implanted pacemaker or defibrillator
* History of pericarditis
* Congenital heart disease
* Coagulopathy or bleeding disorders
* Contraindications to oral anticoagulation
* Contraindications to CT or MRI
* Pregnancy or breastfeeding
* Body Mass Index >30
* History of organ transplantation
* Severe pulmonary disease
* Estimated Glomerular Filtration Rate <30 mL/min/1.73 m²
* Active malignancy
* Significant infection
* Life expectancy <1 year
* Psychiatric disorders preventing study participation
* Refusal or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation | 12 months post-procedure
  Any symptomatic or asymptomatic episode of atrial fibrillation lasting >30 seconds, confirmed by ECG or Holter monitoring.

SECONDARY OUTCOMES:
Intraprocedural bradyarrhythmic episodes | During ablation procedure
  Number of Participants with periprocedural occurrence of bradyarrhythmias lasting >10 seconds that require atropine administration or temporary pacing.
Requirement for intraprocedural cardioversion | During ablation procedure
  Number of Participants with periprocedural need for electrical cardioversion to terminate atrial fibrillation episodes during the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Heart Rhythm Center, Rzeszów, Podkarpackie Voivodeship, Poland